CLINICAL TRIAL: NCT07188051
Title: A 12 Week Clinical Study to Evaluate the Effects of an Eggshell Membrane Dietary Supplement on Elasticity and Skin Hydration Versus Placebo
Brief Title: Ovolux Beauty From Within Trial#2
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: ESM Technologies, LLC (Industry)
Collaborators: Princeton Consumer Research Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: STNCLI1Q
Record Dates: First submitted 2025-09-10; First posted 2025-09-23 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Skin Sagging; Skin Wrinkling; Skin Dryness
Keywords: ovolux; eggshell membrane; beauty; skin elasticity; wrinkles; hair; fingernails

STUDY DESIGN:
Intervention Model Description: Single-center, randomized, double-blinded, placebo controlled design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Active intervention (Ovolux)
  Interventions: Dietary Supplement: Ovolux brand eggshell membrane powder
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ovolux brand eggshell membrane powder — Unhydrolyzed eggshell membrane powder
  Arms: Active
Dietary Supplement: Placebo — psyllium husk fiber powder
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness of an eggshell membrane dietary supplement (Ovolux brand) in supporting beauty from within.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the dietary supplement, Ovolux brand eggshell membrane, versus a placebo control for potential effects on facial skin elasticity, hydration, and wrinkles, and hair attributes using bioinstrumentation (Corneometer, Cutometer), imaging (VISIA CR Imaging, HairMetrix analysis) and subjective evaluation of hair, nail and facial skin condition over 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to read, understand, and provide written Informed Consent and Photo Release.
* Participant is a healthy female or male, aged 35 through 65 years (inclusive).
* Participant is willing and able to swallow capsules.
* Participant has self-perceived facial wrinkles and facial sagging skin.
* Participant is seeking improvements to hair and nails such as hair growth and thickness and nail strength and appearance.
* Participant agrees to keep their hair at least 3 inches long.
* Participant is willing to comply with all study procedures and attend all study visits.
* Participant agrees not to have any hair cosmetic procedures such as relaxers or perms, etc. while on the study. Coloring/dyeing is permitted if part of the participant's regular routine and this routine is maintained during the study.
* Participant is willing to forego taking any hair, nail or skin supplements or using/applying any other hair, nail or skin products on their hair/scalp, nails or face that promote nail or hair growth or are collagen boosting for the duration of the study.
* Participant is willing to discontinue any hair or nail or collagen boosting dietary or nutritional supplements two weeks before the onset of the study and for the study duration. Dietary supplements such as a general multi-vitamin, vitamins A, C or D, iron or calcium are acceptable.
* Participant agrees not to wet their face or consume hot or cold or caffeine containing foods or beverages within 2 hours of all visits.
* Participant reviewed the ingredient list for the test article (dietary supplement) and the placebo and, to the best of their knowledge, confirmed they have no sensitivity or allergy to the ingredients.
* Females of child bearing potential must agree to use an adequate method of birth control, which include: systemic birth control (must have been on the same type of systemic birth control for at least 3 months prior starting the study and must not change the type of birth control during the study); diaphragm with spermicide, condom with spermicide; IUD (hormonal or copper); Vasectomized partner; bilateral tubal ligation; or Abstinence. Females who are post-menopausal (absence of menses for at least 1 year), have had a hysterectomy or have had a bilateral oophorectomy do not need any additional birth control are considered to be not of childbearing potential; (Confirmed by verbal response only).

Exclusion Criteria:

* Participant is allergic to eggs or egg proteins.
* Participant is a smoker.
* Participant has a current skin disease on or near the scalp (e.g., eczema, psoriasis) or anywhere else on the body.
* Participant has any allergies or sensitivities to any dietary or nutritional supplements or their ingredients.
* Participant has artificial nails (press-on, glue-on, gel, acrylic, etc.). Nail polish is permitted if part of regular nail routine and if this routine is maintained during the study.
* Participation in another supplement study in the past 30 days.
* Participant has dreads or weaves.
* Participant has had any chemical hair procedure (used relaxers, perms, etc.) in the last 8 weeks.
* Participant has dyed their hair within the last 3 days.
* Participant has a diagnosed hair loss disorder such as alopecia areata, scarring alopecia, and/or androgenetic alopecia and/or pattern baldness.
* Participant is taking or using any medications or supplements (over the counter or prescription, topical or oral) for hair growth such as minoxidil, finasteride, dutasteride, spironolactone, collagen, amino acids, keratin, biotin, rosemary oil, corticosteroid injections, etc. or treatments for hair growth such as laser treatment or supplements for nails or skin.
* Participant is under treatment by a medical professional for a hair/scalp, nail or skin condition.
* Participant has any concomitant skin diseases of the scalp or skin such as atopic dermatitis, seborrheic dermatitis, psoriasis, eczema, tinea capitis, etc. or irritation such as rash, sores, etc. on the scalp.
* Participant has an infestation on the scalp such as lice.
* Female Only: Participant is pregnant, planning to become pregnant during the course of the study or nursing (self-reported).
* Participant has been diagnosed with chronic skin allergies.
* Current use of OTC pain medication ingested in quantities exceeding label use.
* Participant has been diagnosed with any type of cancer especially skin cancer within the past 12 months or treated for cancer in the last 5 years.
* Participant is routinely using any anti-inflammatories, and/or antihistamines.
* Participant has a history of any chronic diseases such as insulin dependent diabetes, HIV/AIDS, etc.
* Participant has any medical condition or is taking a medication that would compromise the safety of the participant or preclude participation in the study per the Principal Investigator.
* Participant is currently participating in another clinical trial involving the skin, scalp or hair or nails.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
Change in Skin Elasticity | Baseline, Week 4, Week 8, and Week 12
  Measurement of facial skin elasticity parameters (R0, R2, R5, R6 and R9) via Cutometer® to determine if it improves or worsens

SECONDARY OUTCOMES:
Change in Skin Hydration | Baseline, Week 4, Week 8, and Week 12
  Measurement of facial skin hydration via Corneometer® to determine if it improves or worsens
Change in Hair Thickness/Density | Baseline, Week 12
  Trichoscopy to evaluate hair attributes using D200evo Dermatoscope with HairMetrix® to determine if thickness/density improves or worsens
Change in Skin Wrinkles | Baseline and Week 12
  VISIA images will be collected for analysis of facial wrinkles to determine if wrinkling improves or worsens
Participant Self-Assessment Questionnaires | Baseline, Week 4, Week 8, and Week 12
  Self-Assessment Questionnaires for skin, hair, & fingernail quality completed by participants. Each scale ranges from zero (poor) to ten (excellent). Higher scores equate to a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Princeton Consumer Research Corp., Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No